CLINICAL TRIAL: NCT02474875
Title: Explain Pain in Fibromyalgia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Collaborators: Universidad Rey Juan Carlos (Other); University of Alcala (Other); University of Valencia (Other)
Responsible Party: Principal Investigator, J.J. Amer-Cuenca, Head of Department, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEI14 / 008
Record Dates: First submitted 2015-06-12; First posted 2015-06-18 (Estimated); Last update posted 2018-10-01 (Actual); Status verified 2018-09

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia; Patient education; Central sensitization
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Educational program Control Group (Active Comparator): 6 group sessions: 1h/session - 1 session/week - 6 weeks 4 first sessions: relaxation exercises 2 last sessions: talk about medical issues (drugs, nutrition, importance of sleep...)
  Interventions: Other: Educational program
- Educational program High Dose Group (Experimental): 6 group sessions: 1h/session - 1 session/week - 6 weeks 6 sessions: 45 minutes of educational sessions about the neurophysiology of pain + 15 minutes of relaxation exercises
  Interventions: Other: Educational program
- Educational program Diluted Low Dose Group (Experimental): 6 group sessions: 1h/session - 1 session/week - 6 weeks 6 sessions: 45 minutes of educational sessions about the neurophysiology of pain + 15 minutes of relaxation exercises
  Interventions: Other: Educational program
- Educational program Concentrated Low Dose Group (Experimental): 6 group sessions: 1h/session - 1 session/week - 6 weeks 4 first sessions: relaxation exercises 2 last sessions: educational sessions about the neurophysiology of pain
  Interventions: Other: Educational program

INTERVENTIONS:
Other: Educational program — Patients in experimental groups will receive different educational sessions (contents and duration)

SUMMARY:
Education of pain physiology is described as an educational session or sessions describing the neurobiology and neurophysiology of pain, and pain processing by the nervous system. There is compelling evidence that an educational strategy addressing neurophysiology and neurobiology of pain can have a positive effect on pain, disability, catastrophization, and physical performance in chronic musculoskeletal pain disorders. Although pain physiology education has been studied in patients with chronic low back pain, chronic whiplash, and chronic fatigue syndrome in combination with widespread pain, studies in fibromyalgia (FM) are limited to a 2013 study with limited results.

The investigators propose a study with a higher dose of education of pain physiology (i.e. a higher number of educational sessions and total education time) to study if this generates a larger treatment effect in patients with fibromyalgia.

ELIGIBILITY:
Inclusion Criteria:

* American College of Rheumatology classification criteria for FM, both 1990 and 2010
* Reported average pain intensity ≥ 4 on a 0 to 10 cm visual analogue scale based on 1 week of daily pain diaries
* On stable doses of medications for FM ≥ 4 weeks

Exclusion Criteria:

* Suffer from an inflammatory rheumatic conditions
* Have a planned elective surgery during the study period
* Have ongoing unresolved disability claims
* Experience symptoms of bipolar disorder, major depressive disorder, panic disorder, or psychosis
* Do not speak Spanish fluently

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analog Scale | Baseline - 6 weeks - 3 months
  On this continuous, horizontal scale used, where 0 is ''no pain" and 100 is ''worst possible pain" (0-100 mm line), subjects will be asked to mark the line with a cross somewhere between both extremes that best reflect their sensation

SECONDARY OUTCOMES:
Change in Fibromyalgia Impact Questionnaire | Baseline - 6 weeks - 3 months
  A validated self-reported questionnaire developed for FM (scores range from 0 to 100, average FM patients score about 50 and severely affected patients score >70) wich measures multidimensional function/health-related quality of life.
Change in Pressure Pain Threshold | Baseline - 6 weeks - 3 months
  The Pressure Pain Threshold (PPT) is defined as the lowest pressure that, using standardized testing conditions, needs to be applied in order to cause the slightest sensation of pain. It is a reliable and widely used measure. PPTs will be the average intensity of three consecutive measurements, applied every 30 seconds, measured using an analogue Wagner algometer (Wagner Instruments, Greenwich, CT) fitted with a 1 cm2 pressure, with an approximate rate of pressure increase of 1 Kg/s.
Change in Medical Outcomes Study Short Form 36 (SF-36) | Baseline - 6 weeks - 3 months
  The Physical Component Summary score of the Medical Outcomes Study Short Form 36 [SF-36] will be used. More than 10% improvement in SF-36 physical function has been identified as a responder-to-treatment definition for FM clinical trials
Change in Patient Global Impression of Change Scale | Baseline - 6 weeks - 3 months
  The patient global impression of change scale (PGIC) is recommended for evaluating participant ratings of overall improvement in pain treatment trials. The PGIC uses a 7-point Likert scale that varies from 1 "very much improved" to 7 "very much worse" to quantify patient global response to treatment and have been previously used in FM treatment trials.
Change in Depression subscale of the Hospital Anxiety and Depression Scale | Baseline - 6 weeks - 3 months
  The Depression subscale of the Hospital Anxiety and Depression Scale (HADS-D) includes 7 items to assess depressive symptoms, with each item answered on a four-point (0 to 3) scale so that possible scores range from 0 to 21 with higher scores indicating more severe symptoms. An analysis of data from three pregabalin FM trials supports diagnostic validity of the HADS by showing that, using a standard cutoff score of ≥11 on the HADS-D to identify patients with major depressive disorder
Change in Fatigue Severity Scale | Baseline - 6 weeks - 3 months
  The Fatigue Severity Scale (FSS)20 is a 9-item unidimensional measure of fatigue that has been demonstrated to be valid and reliabile in FM patients. The FSS measures fatigue by quantifying the impact of fatigue on specific types of functioning. Each item is scored on a 7-point rating scale, and the FSS score is derived by averaging all items to yield a score from 1 to 7 with higher scores indicating more severe fatigue symptoms.
Change in Jenkins Sleep Scale | Baseline - 6 weeks - 3 months
  The Jenkins Sleep Scale (JSS) is a 4-item self-report questionnaire designed to measure how often a subject has experienced sleep problems in the past month and has been studied in FM patients and found to be valid, reliable, and able to detect change after treatment. JSS items evaluate trouble falling asleep, staying asleep, waking up several times, and awakening unrefreshed with each item scored on a 5-point Likert scale from 0 = "not at all" to 5 = "22-31 days." Scores vary from 0 to 20 with higher scores indicating more frequent sleep problems.
Change in Manual Tender Point Survey | Baseline - 6 weeks - 3 months
  The Manual Tender Point Survey (MTPS) is a standardized approach to performing the tender point exam in which FM patients rate pain severity upon digital palpation of each tender point on a verbal 11 point number rating scale. Pain severity ratings from the 18 tender points are averaged to yield a Fibromyalgia Intensity Score (FIS) that varies from 0 to 10 with higher scores indicating more severe tenderness. Change in the severity of pain at tender point sites has been shown to be a better measure of tenderness than change in the number of tender points.
Change in Neurophysiology of Pain Test | Baseline - 6 weeks - 3 months
  The Neurophysiology of Pain Test-patient version consists of 19 true-false choice items (scores ranging from 0 to 19, with high scores representing a better knowledge regarding pain neurophysiology). This test evaluates whether patients can understand currently accurate information about the neurophysiology of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Juan J. Amer-Cuenca, Study Director — Head of Physical Therapy Department
Locations (4):
- Spain (4):
  - Unviversidad de Alcalá, Alcalá de Henares
  - Universidad Rey Juan Carlos, Alcorcón
  - Universidad CEU Cardenal Herrera, Valencia
  - Universidad de Valencia, Valencia

REFERENCES:
- [Background] Van Oosterwijck J, Meeus M, Paul L, De Schryver M, Pascal A, Lambrecht L, Nijs J. Pain physiology education improves health status and endogenous pain inhibition in fibromyalgia: a double-blind randomized controlled trial. Clin J Pain. 2013 Oct;29(10):873-82. doi: 10.1097/AJP.0b013e31827c7a7d. PMID 23370076
- [Background] van Ittersum MW, van Wilgen CP, Groothoff JW, van der Schans CP. Is appreciation of written education about pain neurophysiology related to changes in illness perceptions and health status in patients with fibromyalgia? Patient Educ Couns. 2011 Nov;85(2):269-74. doi: 10.1016/j.pec.2010.09.006. Epub 2010 Sep 29. PMID 20880654
- [Background] Boomershine CS. A comprehensive evaluation of standardized assessment tools in the diagnosis of fibromyalgia and in the assessment of fibromyalgia severity. Pain Res Treat. 2012;2012:653714. doi: 10.1155/2012/653714. Epub 2011 Oct 10. PMID 22110942
- [Background] Bowering KJ, O'Connell NE, Tabor A, Catley MJ, Leake HB, Moseley GL, Stanton TR. The effects of graded motor imagery and its components on chronic pain: a systematic review and meta-analysis. J Pain. 2013 Jan;14(1):3-13. doi: 10.1016/j.jpain.2012.09.007. Epub 2012 Nov 15. PMID 23158879